CLINICAL TRIAL: NCT02060292
Title: Novel Vascular Manifestations of Chronic Obstructive Pulmonary Disease
Acronym: NOVASC COPD
Status: Completed | Type: Observational
Sponsor: North Bristol NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 3251
Record Dates: First submitted 2013-11-29; First posted 2014-02-12 (Estimated); Last update posted 2018-06-28 (Actual); Status verified 2018-06

CONDITIONS: COPD
Keywords: COPD; Cognitive Function; MRI Brain; Aortic Stiffness; Cerebrovascular disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Cerebrovascular Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD: Stable, Non hypoxaemic, without history of vascular disease
- Healthy smokers: Age matched, smokers without COPD

SUMMARY:
Cognitive impairment is a known consequence of cerebral small-vessel disease. Moderate to severe cognitive impairment has been shown in up to 60% of certain individuals with COPD and is likely to profoundly influence an individual's ability to manage their disease.

In addition to cerebral small vessel damage and cognitive dysfunction, other organs such as the heart, kidneys, and retina are likely to be susceptible to small-vessel damage in COPD. Several large population studies have shown that COPD is a significant independent risk factor for myocardial infarction, with the effect most marked in early, mild disease.

We propose to compare non-invasive MR brain imaging of white matter microstructure (diffusion tensor), cerebral perfusion (arterial spin labelling) and accumulated cerebral small vessel disease (cerebral microbleeds), in COPD patients to smokers without COPD. In addition we plan to explore mechanisms of cerebral small vessel disease in COPD by looking for associations between arterial stiffness, end organ vascular damage and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects must give their signed and dated written informed consent
2. Subjects must be aged >40 and ≤ 85
3. Subjects with a smoking history > 10 pack years.
4. COPD group: Subjects with a FEV/FVC <70%

Exclusion Criteria:

1. Resting oxygen saturations <92% on room air.
2. Long term oxygen therapy
3. Recent exacerbation of COPD (4 weeks)
4. Ischaemic heart disease
5. Cerebrovascular disease
6. Uncontrolled hypertension
7. Diabetes mellitus
8. Hepatic failure
9. Neurological disease
10. Non-cured tumours
11. Obstructive sleep apnoea
12. Current of past alcohol/drug abuse
13. Known history of dementia
14. Visual or hearing impairment that precludes neuropsychological assessment
15. Neuropsychological tests undertaken outside the study
16. Pregnant women or women who are lactating
17. Known alpha 1 anti-trypsin deficiency as a cause of their COPD
18. History of psychiatric disorders, or other conditions that will impact on the validity of their consent or interfere with compliance to perform study procedures.
19. Contra indication to MRI scanning -

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Stable COPD
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2014-04; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Fractional Anisotropy | upto 4 weeks
  MRI Diffusion Imaging - measure of cerebral white matter microstructure

SECONDARY OUTCOMES:
Aortic Pulse Wave Velocity | upto 4 weeks
  Aortic stiffness
MRI Cerebral Perfusion - ASL | upto 4 weeks
Cerebral Microbleeds | upto 4 weeks
Cognitive Function | upto 4 weeks
  Montreal Cognitive Assessment
Cardiac MRI | upto 4 weeks
  LV & RV Mass
FEV1 % predicted | upto 4 weeks
Arterial Oxygen Saturation | upto 4 weeks
Retinal Photography | upto 4 weeks
  Retinal Arterial Narrowing
Micro-albuminuria | upto 4 weeks
  Spot urine albumin sample mg/l (milligram albumin per litre of urine)
Health Status | upto 4 weeks
  COPD Assessment Test (CAT score) 0-40

OTHER OUTCOMES:
Serum Inflammatory Markers | upto 4 weeks
  Fibrinogen, C reacive Protein, IL-6

CONTACTS AND LOCATIONS:
Overall Officials: James W Dodd, MB ChB PhD, Principal Investigator — University of Bristol
Locations (1):
- North Bristol NHS Trust, Bristol, Avon, United Kingdom

REFERENCES:
- [Derived] McKay GJ, McCarter RV, Hogg RE, Higbee DH, Bajaj MK, Burrage DR, Ruickbie S, Baker EH, Jones PW, Dodd JW. Simple non-mydriatic retinal photography is feasible and demonstrates retinal microvascular dilation in Chronic Obstructive Pulmonary Disease (COPD). PLoS One. 2020 Jan 10;15(1):e0227175. doi: 10.1371/journal.pone.0227175. eCollection 2020. PMID 31923188